CLINICAL TRIAL: NCT02754050
Title: Safety and Feasibility of the Tandem Snare Device
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tandem Technologies LTD (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP-001
Record Dates: First submitted 2016-04-19; First posted 2016-04-28 (Estimated); Last update posted 2016-04-28 (Estimated); Status verified 2016-04

CONDITIONS: Polyps
MeSH Terms: conditions — Polyps

ARMS (1):
- Polypectomy (Experimental): When a 6-25mm polyp is identified the Tandem snare will be inserted through the colonoscope, remove and retrieve the polyp.
  Interventions: Device: Tandem Snare

INTERVENTIONS:
Device: Tandem Snare

SUMMARY:
The device is intended to endoscopically transect polyps in the gastrointestinal tract (sessile or pedunculated) using electrocautery. During the same maneuver the polyp is captured, retrieved and submitted for pathological analysis. The Tandem Snare is an intervention tool inserted through the colonoscope for the resection and removal of polyps sized 6 to 25 mm. The Tandem snare utilizes a technology that has the potential to hold the polyp, lift it up, resect and remove it without losing it. This is a feasibility study aiming to demonstrate the safety of the Tandem Snare used for 6-25mm polyps' polypectomy in screening, diagnostic or surveillance colonoscopy.

DETAILED DESCRIPTION:
The colonoscopy procedure is considered the "gold standard" for detecting, diagnosing and treating abnormalities in the colon. Detection and removal of colon polyps is the most significant benefit colonoscopy provides toward the reduction of colorectal cancer mortality and morbidity. The Tandem Snare is an intervention tool inserted through the colonoscope for the resection and removal of polyps sized 6 to 25 mm. The Tandem snare utilizes a technology that has the potential to hold the polyp, lift it up, resect and remove it without losing it. The technology may eliminate the repeated bites with the intervention tool or the need to use additional intervention tools such as the net. It may improve visual perception for resecting the polyp without losing it while removing from the colon. Consequently it may increase the potential for complete polypectomy and reduce intervention time and repetitions, polyp lost, risks and cost. This is a feasibility study aiming to demonstrate the safety of the Tandem Snare used for 6-25mm polyps' polypectomy in screening, diagnostic or surveillance colonoscopy.

ELIGIBILITY:
Inclusion Criteria:

1. Adults > 18 Years
2. Subjects have been scheduled for colonoscopy
3. Subject has signed the informed consent

Exclusion Criteria:

1. Suspected or known active Inflammatory Bowel Disease (IBD)
2. Coagulopathy or thrombocytopenia.
3. Taking dual anti platelet therapy or anti coagulants.
4. Bowel preparation is deemed poor by colonoscopist.
5. Subjects with known or detected (during colonoscopy) moderate/severe diverticular disease.
6. History of familial polyposis (FAP).
7. History of prior surgery to colon and/or rectum.
8. ASA ≥ IV.
9. Pregnancy (as stated by patient).
10. Subjects with altered mental status/inability to provide informed consent.
11. Patients who have participated in another interventional clinical study in the last month.
12. Subject under a condition which in the investigators opinion may put the subject at significant risk, confound study results, or interfere significantly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2016-09; Primary Completion 2018-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Device related major adverse events | 7 days
  Device related major adverse events include death, major bleeding or perforation)
Technical success of the Tandem Snare. | 1 day
  The primary feasibility assessment will be encountered as success if the Tandem Snare was inserted through the working channel, cut the polyp and the device was successfully removed from the working channel.

SECONDARY OUTCOMES:
Retrieval rate of the polyps that have been cut by the Tandem Snare. | 1 day
  The secondary performance assessment will be based on data from all polyps which were resected by the Tandem Snare. Retrieval of the resected polyp will be encountered as success,